CLINICAL TRIAL: NCT00263497
Title: Immediate Temporary Prosthesis Fitting in Traumatic Trans-tibial Amputation: a Controlled Clinical Study in Rural Cambodia
Brief Title: Temporary Prosthesis in Traumatic Below-knee Amputation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No update for several year, confermed ended by Odd Edvardsen i march 2020.
Sponsor: University Hospital of North Norway (Other)
Collaborators: Medical University of Joenkoeping, Sweden (Other); NCHADS - Ministry of Health of Cambodia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KHM1030375
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Transtibial Amputation
Keywords: Postinjury chronic pain; Transtibial amputation; Physical rehabilitation; Immediate temporary prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Temporary tuber-ischii bearing prosthesis — Tuber ischii-bearing holster is connected by hinged metal bars to foot device to enable immediate postoperative mobilization of transtibial amputees. No other medical interventions or pharmaceutical treatment.

SUMMARY:
Most trauma survivors in low-income countries develop post-injury chronic pain syndromes. Normally traumatic amputees have to wait 4-6 months for definitive prosthesis fitting. The actual study aims at reducing post-injury chronic pain and improving function by immediate temporary prosthesis fitting after surgery.

DETAILED DESCRIPTION:
Background: Previous studies document that 75% of traumatic amputees in low-income countries develop incapacitating chronic pain syndromes. With the present level of rehabilitation service, amputees have to wait 4-6 months for postoperative prosthesis fitting.

Hypothesis: Immediate postoperative prosthesis fitting reduce chronic pain and improves function in trans-tibial amputees.

Reference population: Traumatic amputees living in low-income and low-resource communities.

Study population: Adult patients with trans-tibial amputations in rural districts of Battambang Province, Cambodia.

Study design: A semi-cross over controlled study. Supplement:longitudinal qualitative studies of subsets.

Main variables for quantitative study:

* Outcome indicators:Self-rated pain (VAS). Self-rated function (VAS). Pain (clinical exam). Gait analysis.
* Variables: Preinjury morbidity and socioeconomical status. Injury severity (RTS, ISS). Prehospital and hospital analgesia. Postoperative infection. Amputation stump quality (clinical rating).

Sampling: Given test power =0.8, significance level =0.05, sequential analysis of results, an estimate of 15 patients will be included in each study group. The sample may be modified due to sequential analysis (see below).

Intervention: A mobile rural workshop takes molds and adapt temporary tuber-ischii bearing prosthesis made of local materials. The prosthesis is fitted at the time of amputation wound closure (5 - 15 days post-injury), and patients mobilized on walking aids. Control group patients comprise of transtibial amputees managed at neighboring hospitals not being served by the actual rehab workshop. Control patients leave hospital with walking aids without prosthesis. Data are gathered by rehab team (surgeon and prosthesis technician) at point zero, 1 month postoperation, 3 months postoperation. End-point for evaluation is 6 months post-op. Patients decide freely to cross-over on pain indications.

Statistical analysis: Sequential design with positive and negative stopping rules. Outcome variables at end-point are reported for groups of 3 patients to statistician(Prof. Stig Larsen, University of Oslo) who gives stop orders.

Ethical considerations: If ITP proves favorable, the study results will be used to expand the rural rehab service to include control districts as well. This makes the use of control groups in the actual study legitimate. Also optional cross-over prevents against inflicting unnecessary discomfort in study patients. The study is approved by the local health authorities and Norwegian Committee for Research Ethics. The system for data filing and protection is approved by Norwegian Social Science Data Services, Bergen.

Publication: Authorship will be set according to Vancouver regulations.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic transtibial amputation

Exclusion Criteria:

* Double amputation

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Pain: Patient-rated | 1, 3, and 6 months postinjury
Pain: clinical exam rated | 1, 3, and 6 months post-injury
Function: patient-rated | 1, 3, and 6 months post-injury
Function: gait analysis | 1, 3, and 6 months post-injury

SECONDARY OUTCOMES:
Qualitative longitudinal study of subsets | 1, 3, and 6 months post-injury

CONTACTS AND LOCATIONS:
Overall Officials: Bjoern Karlsson, Rehab Ing, Principal Investigator — TMC, University Hospital Northern Norway
Locations (1):
- Trauma Care Foundation Cambodia, Battambang, Cambodia